CLINICAL TRIAL: NCT02936167
Title: Comparison of Ringer Lactate and Isotonic Acetate Solution as Maintenance Fluids in Children Undergoing Elective Laparoscopic Surgery
Brief Title: Comparison of Ringer Lactate and Isotonic Acetate Solution as Perioperative Maintenance Fluid for Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, KARTHIK RAM A, Junior Resident,Dept. of Anaesthesia and Intensive Care ,pgimer, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: NK/2181/MD/11192-93
Record Dates: First submitted 2016-10-12; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Hyponatremia
Keywords: Ringer Lactate; Plasmalyte; Perioperative Period
MeSH Terms: conditions — Hyponatremia | interventions — Ringer's Lactate; Plasmalyte A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ringer Lactate (Experimental): fluid
  Interventions: Biological: Ringer Lactate
- Plasmalyte (Experimental): fluid
  Interventions: Biological: Plasmalyte

INTERVENTIONS:
Biological: Ringer Lactate
  Arms: Ringer Lactate
Biological: Plasmalyte
  Arms: Plasmalyte

SUMMARY:
In children fluids are supplemented during surgery to provide volume, to maintain blood glucose levels, electrolyte balance and to meet the ongoing fluid losses during surgery. Fluid replacement during surgery since decades has been based on the Holliday and Segar method.These authors proposed that water maintenance in children includes: 100 millilitre (ml)/100 kilocalorie (kcal) for the first 10 kg of body weight, 50mL/100 kcal for 11-20 kg and 20mL/100 kcal for every kilogram of body weight above 20 kg. The maintenance electrolyte requirements of 3 mEq/100 kcal for sodium and 2 mEq/100 kcal for potassium per day, were based upon the electrolyte composition of breast and cow's milk. Based on these recommendations hypotonic fluid (0.45% saline) was considered as the ideal fluid for maintenance in children undergoing surgery.

Since the past many years there have been many documented cases of hyponatremia after administration of hypotonic fluids with potential for serious neurological injury in this group of patients.The use of Holliday and Segar's formula to calculate the maintenance fluid regimen in postoperative children leads to an overestimation of the volume of fluid needed, as there is a low urine output in this period. The postoperative period is at risk for non-osmotic secretion of anti-diuretic hormone (ADH), which reduces the ability of kidney to excrete free water and carries risk for development of hyponatraemia.Authors in favour of hypotonic solutions feel that hyponatremia results from excessive volume of fluid and isotonic solutions have risk of hypernatremia, interstitial fluid overload, excessive sodium excretion, and hyperchloremic metabolic acidosis.

Based on the increased incidence of hyponatremia in children undergoing surgery, the paediatric anaesthesia societies [Society of Paediatric Anesthesia (SPA), Paediatric Anaesthesia Society of Great Britain and European society of Paediatric Anesthesia (ESPA)] put forward guidelines for the type and amount of fluid to be administered during surgery.Since then normal saline is the commonly used fluid during the perioperative period.However recent studies have shown that the use of normal saline is associated with development of hyperchloremic metabolic acidosis and poor outcome.

Ringer lactate (RL) is a commonly used intravenous fluid during surgery and has been found to have decreased possibility of producing hyponatremia although it is a slightly hypotonic solution.Plasmalyte is an isotonic fluid which has been shown to maintain electrolyte balance and prevent hyponatremia as well as hyperchloremic acidosis in adult population.However plasmalyte has been less frequently used in paediatric population.Therefore this study is planned with the aim of comparing intravenous fluids, ringer lactate and plasmalyte in the perioperative period regarding the incidence of hyponatremia produced by these solutions, their effect on electrolytes and blood gases in children undergoing elective surgery.

DETAILED DESCRIPTION:
Fluid therapy is aimed to compensate for fasting which is required for surgery, to meet the ongoing fluid losses and to maintain electrolyte balance during surgery. Fluid deficit of a healthy child who is not fed parenterally may be estimated by multiplying hourly maintenance requirement for fluid by number of hours since the child's last oral intake (50% of deficit + maintenance in first hour, 25% of deficit + maintenance in second hour). Maintenance fluid therapy represents the volume of fluids and amount of electrolytes and glucose needed to replace anticipated physiological losses from breath, sweat and urine and to prevent hypoglycaemia. This maintains homeostasis while an individual is unable to control his/her own fluid intake while being operated. Replacement fluid represents the volume of fluid given to replace the volume lost during the surgical procedure. For 50 years, this therapy was based on Holliday and Segar's formula.

In 1957, Malcolm Holliday and William Segar published fluid management guide-lines for hospitalized children, which proposed to match children's water and electrolyte requirements on a weight-based calculation using: 100 ml/100 kcal for the first 10 kg of body weight, 50 ml/100 kcal for 11-20 kg and 20 ml/100 kcal for every kilogram of body weight above 20 kg. Their proposed maintenance electrolyte requirements of 3 meq/100 kcal of sodium (Na) per day and 2 meq/100 kcal of potassium (K) per day, were based upon the electrolyte composition of breast and cow's milk.

Once applied, these recommendations identified hypotonic fluid as the ideal maintenance fluid choice in hospitalized children, leading to the widespread use of 0.225% and 0.45% saline in this population. However, the widely used recommendations of Holliday and Segar did not consider the changing fluid and electrolyte requirements of a sick or postoperative child. Hypotonic fluid with a low sodium content (77 meq/l) and high percentage of electrolyte free water (78% EFW) can cause dilutional hyponatremia.Along with this, non-osmotic stimuli of anti-diuretic hormone (ADH) secretion in postoperative period makes the patient more vulnerable to hyponatremia. The primary stimulus for ADH release is an increase in osmolality however, many non-osmotic stimuli like nausea have also been identified as a potent non-osmotic stimulus for ADH release.Non osmotic causes of ADH release are broadly divided into hemodynamic and non-hemodynamic stimuli for its release. Hypovolemia, hypotension, hypoalbuminemia, congenital heart failure are some hemodynamic causes of non-osmotic secretion of ADH. Pneumonia, bronchitis, hypoxia, meningitis and brain tumour are some of the non-hemodynamic causes of ADH release.

Anti-diuretic hormone (ADH), is a neurophysial hormone which is synthesised in the supraoptic nuclei of the hypothalamus and released from the posterior pituitary gland. It binds to vasopressin V2 receptor in the basolateral membrane of the collecting duct, which leads to the insertion of aquaporin-2 receptors for retaining water in the body. By retaining water and decreasing urine output it increases the electrolyte free water in vascular compartment causing hyponatremia.Hyponatremia leads to hypotonicity of extracellular fluid (ECF) resulting in movement of water into intracellular space hence cell swells and cerebral edema occurs.Clinical presentation of acute hyponatremia (decrease in Na over ≤48 hours to <135meq/L) includes headache, lethargy and seizures, and potentially even respiratory and cardiac arrest secondary to brain stem herniation.2,3 These outcomes are more likely to be seen with severe acute hyponatremia (Na <130 mmol/L) and because of their higher brain/intracranial volume ratio, children are at increased risk for these sequelae compared with adults.Several studies have consistently showed that postoperative patients have an increased risk of developing hyponatremia.The incidence of hyponatremia after administration of hypotonic solutions varies from 11 to 31%.

Arieff et al, conducted a prospective clinical case study of 16 children and reviewed 24,412 children admitted for surgery. The main objective was to find out whether hyponatremia causes permanent brain damage or not. Over a period of 6 years, 16 children admitted in 5 tertiary hospitals and 9 community hospitals developed hyponatremia within 5 days of admission. At admission the sodium levels were 138 mmol/l. Patients became progressively lethargic, complained of nausea and vomiting after 2 hours of hypotonic fluid infusion. After 37 hours serum sodium was 115 mmol/l and urine osmolality was 676 mmol/kg. Among 16 patients, one was mentally retarded, 10 died and 5 were in permanent vegetative state. Four patients treated with IV sodium chloride (154 mmol/l and 512 mmol/l) showed an increase in sodium level from 108 to 138 mmol/l in 44 hours. Among 24,412 patients 83 patients developed postoperative hyponatremia out of which 7 died.

Grissenger, published case reports of hyponatremia and death in two healthy children who were administered plain dextrose and hypotonic saline after surgery. First child underwent tonsillectomy and adenoidectomy. The child was given maintenance fluid of 5% Dextrose 200ml/hr instead of 75ml/hr due to calculation error. The child vomited several times, became lethargic and threw seizures. The secondchild underwent repair of coarctation of aorta and was given IV frusemide 1mg/hr as the child's urine output was low. On postoperative day-2 child developed hyponatremia and sodium chloride infusion was started as per physician's order. In the morning the child became less responsive and by afternoon he developed seizures and vomiting. In both cases by the time the intensivist could recognize hyponatremia and start treatment, the child became unresponsive to pain stimuli. Despite intubation, ventilatory support, aggressive sodium correction and treatment of cerebral edema both the children died.

Eulmesekianet al, conducted a prospective observational study on postoperative patients admitted in paediatric intensive care unit to establish incidence and factors associated with hospital acquired hyponatremia. A total of 81 patients having serum sodium in normal range (136-146 mmol/l) and requiring IV fluid in the post-operative period were included in the study. The incidence of hospital-acquired hyponatremia at 12 hrs was 21% [95% CI (3.7-38.3)], at 24 hrs it was 31% [95% Confidence interval (CI)(11.4-50.6)]. At 12 hrs, relative risk of developing hyponatremia was 11.55 (95% CI [ 2.99-44.63]; p =0.0004) for Na loss of >0.5 mmol/kg/hr, RR=10 (95% CI, 2.55-39.15; p=0.0009) for a negative Na balance of >0.3 mmol/kg/hr, and RR=4.25 (95% CI,1.99-9.08; p=0.0002) for a urine output >3.4 mL/kg/hr. At 24 hrs, relative risk for hyponatremia was 3.25 (95% CI [1.2-8.77]; p =0.0201) for a positive fluid balance of > 0.2 mL/kg/hr.

Choong et al, conducted a randomized controlled study involving 258 patients aged 6 months to 16 yrs of age with expected postoperative stay of >24hrs. Patients with uncorrected plasma sodium level, abnormal ADH secretion, recent diuretic use, on total parenteral nutrition were excluded from study. Patients were randomized into hypotonic perioperative maintainence solution(PMS) (n=130) or isotonic PMS (n=128) group by a computer generated randomization sequence. The primary outcome was hyponatremia occurring during study intervention and secondary outcomes were severe hyponatremia, hypernatremia, and plasma ADH levels. This study showed that the risk of hyponatremia was greater for patients who received hypotonic PMS, compared with isotonic PMS (40.8% vs 22.7%; RR: 1.82 [95% CI: 1.21-2.74]; P=0.004). Eight patients (6.2%) developed severe hyponatremia following hypotonic PMS, compared with 1 patient (0.8%) in the isotonic PMS group (RR: 7.21 [95% CI:0.93-55.83]; P =0.059). The risk of hypernatremia was not significantly different between the 2 groups.

Saba et al, conducted a randomized controlled trial involving 59 children aged 3 months to 18 years of age. They were randomized into isotonic and hypotonic groups. The study showed that 24% of the patients in the 0.45% saline group experienced a drop in serum [Na], compared with 19% of those in the 0.9% saline group (p = 0.7). The lowest exit Na (133 mmol/L) and maximum rate of fall (-0.52 mmol/L/h) were in a surgical patient receiving 0.45% saline. This patient had 380 ml of oral fluid intake during the study interval. The second lowest exit Na (135 mmol/L) and next fastest rate of fall (-0.40 mmol/L/h) were in a medical patient receiving 0.9% saline; oral intake was 82 ml. There were no adverse events. No participant developed hypertension.

Neville et al, conducted a prospective randomized study involving 124 children aged 6 months to 15 years admitted for surgery. They received isotonic or hypotonic fluid at 100% or 50% maintenance rate. Plasma electrolytes, osmolality and ADH at induction of anesthesia were compared with values at 8 hours (T8), and 24 hours (T24) after surgery.Blood glucose and ketones were measured every 4 hours. Electrolytes and osmolality were measured in urine samples. The study showed that plasma sodium concentrations fell in both N/2 groups at T8 (100%: -1.5mmol/L, 50%: -1.9 mmol/L; [P < 0.01]) with hyponatremia more common than in the NS groups at T8 (30% vs 10%;[P = 0.02]) but not T24. Median plasma antidiuretic hormone concentration increased 2 to 4 fold during surgery (P <0.001) and only reattained levels at induction of anesthesia by T24 in the N/2 100% group. Two children on 100% developed syndrome of inappropriate ADH secretion (SIADH) (1NS). Fourteen children (23%; 7NS) on 50% maintenance were assessed as dehydrated. Dextrose content was increased in 18 for hypoglycemia or ketosis.

Friedman et al, conducted a randomized controlled trial involving 110 patients aged 1 month to 18 years of age. Patients were randomized into 0.9% saline (isotonic) group and 0.45% saline (hypotonic) group.The primary outcome was to measure mean sodium level at 48 hours.The secondary outcomes were mean sodium level at 24 hours, hyponatremia, hypernatremia, weight gain, edema and hypertension. The mean Na levels in isotonic and hypotonic group were similar. Two of the 56 patients developed hyponatremia in hypotonic group (serum sodium levels of 134meq/l after 24 hours). Mean serum sodium levels at 24 hours did not differ between the groups (140.5 [2.7] vs 139.6 [2.7] meq/l respectively, [95% CI:-0.22 to 2.02 meq/l]; p=0.14. One patient in each group developed hypernatremia with serum sodium levels of 147meq/l at 24 hours. Two patients in each group developed hypertension and 2 patients in the isotonic group developed edema.

Valadaoa et al, conducted a randomized controlled trial involving 57 children aged 1 to 14 years with acute appendicitis and eligible for appendectomy. They were randomized to receive intravenous isotonic or hypotonic maintenance solutions. Samples were collected for measuring electrolytes, urea, creatinine at the start of the infusion, 24 hours and 48 hours after surgery and then analysed. The primary end point of the study was serum sodium levels during the intervention and at the end of 48 hours of the protocol. At admission, 49% patients had moderate hyponatremia (Na=130-135 meq/L) and 51% had normal sodium (Na >136 mEq/L). After 24 hours, 12 patients had hyponatremia of whom 7 had received hypotonic solution. After 48 hours, 17 children had hyponatremia of whom ten had received hypotonic solution. Between the initial Na and final Na levels, there was an increase of 0.9 mEq/L sodium in the isotonic group and of 0.4 mEq/L sodium in hypotonic group. In the group of eight patients with normal initial sodium (>136 mEq/L) and low final sodium (<135 mEq/L) three had received isotonic and five had received hypotonic saline solution with an initial variation of 136 to 140 mEq/L and of 132 to 135 meq/l at 48 h. In the group admitted with low sodium (130-135 mEq/L), nine children remained hyponatremic (132-135 mEq/L) at the end, of whom four had received isotonic solution and five hypotonic solution. Of the 15 patients who had initial hyponatremia (130-135 mEq/L) and normal Na at 48 h (136-140 meq/l) seven received isotonic solution and eight hypotonic solution.

Mc Nab et al, conducted a meta-analysis which included randomized controlled trials comparing isotonic vs hypotonic IV fluids as maintenance fluid in children involving 1109 children aged 3 months to 18 y. The intervention group received isotonic fluid (sodium >125 - 160 meq/l) while the other group received hypotonic fluid (sodium <125 meq/l). The primary outcome of the study was to measure proportion of patients in each treatment group with hyponatremia or hypernatremia at any time point while receiving intravenous fluids. Anti-diuretic hormone level, plasma and urine osmolarity, electrolytes were also measured. A total of 449 patients in the analysis received isotonic fluid, while 521 received hypotonic fluid. Those who received isotonic fluid had substantially lower risk of hyponatraemia (17% versus 34%; RR 0.48; 95% CI 0.38 to 0.60). It was not clear whether there is an increased risk of hypernatraemia when isotonic fluids are used (4% versus 3%; RR 1.24; 95% CI 0.65 to 2.38), although the absolute number of patients developing hypernatraemia was low.

Based on the findings of various studies isotonic fluid like 0.9% normal saline was introduced in clinical practice in paediatric patients undergoing surgery.

Ringer lactate (273 mosm/l) is mildly hypotonic to plasma (294 milliosmol/l) and has been used as maintenance fluid in few studies. These studies showed reduced incidence of hyponatremia and metabolic acidosis when ringer lactate was used as a maintenance fluid.

Zunini et al,retrospectively studied 122 children undergoingcraniofacial surgery. Out of 122 patients 63 received only Normal saline (NS group) whereas 59 received Ringer lactate (RL group). Acid-base balance and electrolytes were measured at 1-2 hrs post-induction (P1) and 2-4 hrs post induction (P2). This study showed that the incidence of metabolic acidosis was 45% (44 patients) in P-1 and 60% (61 patients) in P-2 time period. Acidosis was more frequent in NS group than in the RL group in both periods: 66% and 80% in NS versus 26% and 37% in RL group (P = 0.015 for P-1 and P = 0.027 for P-2). The incidence of severe acidosis (pH <= 7.25) was also larger in those receiving NS (39%) than in those receiving RL (8%). Hyponatremia (Na <135 mmol/L) was observed in 40% (NS) and 26% (RL) of the cases during P-1 and in 52% (NS) and 50% (RL) of the cases during P-2 time period. No statistically significant difference was found in the incidence of hyponatremia between the groups. Overall the incidence of metabolic acidosis and hyponatremia was less in RL group compared to NS group.

Coulthard et al, conducted a randomized controlled trial involving 82 patients undergoing spinal instrumentation, craniotomy for tumor resection or cranial vault remodelling. Children were randomized to receive Hartman's solution with 5% dextrose or 0.45% saline with 5% dextrose. The primary outcome was to measure sodium at 16-18 hours postoperatively. Thirty nine children received Hartman's solution and 40 received hypotonic saline. The result showed mean postoperative plasma sodium levels of children receiving 0.45% saline and 5% dextrose were 1.4 mmol/l (95% CI [0.4 to 2.5]) lower than those receiving Hartmann's and 5% dextrose (p=0.008). In the 0.45% saline group, seven patients (18%) became hyponatraemic (Na <135 mmol/l) at 16-18 postoperatively; in the Hartmann's group no patient became hyponatraemic (p=0.01). No child in either fluid group became hypernatraemic.

Plasmalyte is balanced salt solution with constituents similar to that of plasma, with an osmolality of 294 mosmol/l. In adults, studies using plasmalyte have shown decreased incidence of hyponatremia and metabolic acidosis when compared to hypotonic saline.

McNab et al conducted a randomized controlled double blind study in paediatric population aged 3 months to 18 years of age, comparing plasmalyte and hypotonic saline as maintenance fluid. The patients were randomly assigned into NA-140 and NA-77 group by a computer generated online randomization system. Study investigators, treating clinicians, nurses, and patients were masked to assigned fluid type throughout the study. Eligible patients were started on NA-140 or NA-70 and continued till the maintenance requirement became 50% of standard maintenance rate. When a patient had a surgical procedure before the start of intravenous maintenance fluid, the serum sodium was taken at the end of the procedure and serum electrolytes, urea, creatinine were measured after 6, 24, 48 and 72 h of treatment, until the study fluid was stopped. This study showed that 4% of participants (12 out of 322 ) allocated to Na140 developed hyponatraemia whereas 11% of participants (35 out of 319) developed hyponatremia in Na77 group (odds ratio 0.31,p=0.001). Seven patients developed severe hyponatraemia during the study with little evidence of a difference between the two treatment groups (odds ratio of 0.35, 95% confidence interval of 0.07-1.8; p=0.2). None of these children developed severe hyponatraemia. The occurrence of hypernatraemia was similar in the two groups: 14 (4%) participants developed hypernatraemia in the Na140 group, compared with 18 (6%) in the Na77 group (odds ratio of 0.80, 95% CI of 0.39-1.65,p=0.55).

Since very few studies have been conducted in paediatric population using Ringer Lactate and isotonic acetate solution, this study was planned.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2 - 8 years
* American society of anesthesiologist (ASA) - 1
* Laparoscopic surgical procedure of 2 hours duration requiring IV fluid administration for at least 24 hours

Exclusion Criteria:

* Uncorrected plasma sodium level before surgery
* Diseases which cause abnormal ADH secretion
* Renal and cardiac disease
* Chronic lung disease
* Cranial/thoracic surgery
* Recent loop diuretics use

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
To find out the incidence of hyponatremia and hypernatremia between ringer lactate group and plasmalyte group | 6 months

SECONDARY OUTCOMES:
To find out changes in serum antidiuretic hormone level between Ringer lactate and plasmalyte group | 6 months
To find out changes in urine electrolytes between Ringer lactate and plasmalyte group | 6 months
To find out changes in urine osmolality between Ringer lactate and plasmalyte group | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Neerja Bhardwaj, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] McNab S, Duke T, South M, Babl FE, Lee KJ, Arnup SJ, Young S, Turner H, Davidson A. 140 mmol/L of sodium versus 77 mmol/L of sodium in maintenance intravenous fluid therapy for children in hospital (PIMS): a randomised controlled double-blind trial. Lancet. 2015 Mar 28;385(9974):1190-7. doi: 10.1016/S0140-6736(14)61459-8. Epub 2014 Dec 1. PMID 25472864
- See also: 140 mmol/L of sodium versus 77 mmol/L of sodium in maintenance intravenous fluid therapy for children in hospital (PIMS): a randomised controlled double-blind trial — http://dx.doi.org/10.1016/S0140-6736(14)61459-8